CLINICAL TRIAL: NCT04537884
Title: A Phase 1, Open-Label, Single Ascending Dose Study to Assess the Safety and Tolerability of a Single Intravitreal Injection of UBX1325 in Patients With Diabetic Macular Edema or Neovascular Age-Related Macular Degeneration
Brief Title: Safety and Tolerability Study of UBX1325 in Patients With Diabetic Macular Edema or Neovascular Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBX1325-01
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Macular Edema; Neovascular Age-related Macular Degeneration
Keywords: Retinal disease; Macular edema; Diabetes mellitus; Diabetic macular edema; Neovascular Age-Related Macular Degeneration
MeSH Terms: conditions — Retinal Diseases; Macular Edema; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment with UBX1325 (Experimental): UBX1325, single intravitreal injection, ascending dose
  Interventions: Drug: UBX1325

INTERVENTIONS:
Drug: UBX1325 — Investigational drug intravitreal injection

SUMMARY:
A study to evaluate safety, tolerability, and pharmacokinetics of a single intravitreal injection of UBX1325 in patients diagnosed with diabetic macular edema (DME) or neovascular Age-Related Macular Degeneration.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, first-in-human (FIH), single-ascending dose (SAD) study consisting of approximately 4 cohorts. The total number of patients will be at least 3 per cohort plus 3 additional patients in the maximum tolerated dose (MTD) cohort in order to address the primary objective. Up to an additional 6 nAMD patients will be enrolled in the highest dose cohort. A single dose of UBX1325 will be administered intravitreally and all patients will be followed for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

* nAMD patients who, in the opinion of the Investigator, are inadequately responding to or failed current treatment options.
* Active choroidal neovascularization (CNV) associated with age-related macular degeneration as evidenced on FA and SD-OCT at Day 1, including presence of intraretinal or subretinal fluid.
* BCVA in the study eye (most affected) of 70 Early Treatment Diabetic Retinopathy Study (ETDRS) letters or worse at screening and on Day 1.
* Patients who have the capacity to give informed consent and who are willing and able to comply with all study-related procedures and assessments.

Exclusion Criteria:

* Any ocular/intraocular/periocular infection or inflammation in either eye in the past 4 weeks prior to screening.
* Subretinal hemorrhage with bleeding area ≥4 disc area in the study eye
* Concomitant therapy with anti-VEGF therapies (e.g., Avastin®, Lucentis®, or Eylea®) or previous use of these agents in the study eye within approximately 28 days of study enrollment
* Any retinovascular disease or retinal degeneration other than nAMD in the study eye.
* History of systemic and intraocular steroid use for 6 months prior to Day 1. The use of intravitreal nonbiodegradable steroid implants (ex. Iluvien®, Yutiq®, Retisert®) is prohibited.
* Significant media opacities, including cataract, which might interfere with VA, assessment of toxicity, or fundus imaging.
* Any uncontrolled medical condition that, in the opinion of the investigator, would preclude participation in this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Ocular and systemic safety and tolerability of a single intravitreal injection of UBX1325 evaluated by the incidence of dose limiting toxicities (DLTs) and treatment emergent adverse events (TEAEs) | 24 weeks

SECONDARY OUTCOMES:
Plasma concentration of UBX1325 following a single intravitreal injection | up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Dananberg, MD, Study Chair — UNITY Biotechnology
Locations (8):
- United States (8):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Salehi Retina Institute, Huntington Beach, California
  - MedEye Associates, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - MidWest Eye Institute, Indianapolis, Indiana
  - Houston Eye Associates, Houston, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crespo-Garcia S, Fournier F, Diaz-Marin R, Klier S, Ragusa D, Masaki L, Cagnone G, Blot G, Hafiane I, Dejda A, Rizk R, Juneau R, Buscarlet M, Chorfi S, Patel P, Beltran PJ, Joyal JS, Rezende FA, Hata M, Nguyen A, Sullivan L, Damiano J, Wilson AM, Mallette FA, David NE, Ghosh A, Tsuruda PR, Dananberg J, Sapieha P. Therapeutic targeting of cellular senescence in diabetic macular edema: preclinical and phase 1 trial results. Nat Med. 2024 Feb;30(2):443-454. doi: 10.1038/s41591-024-02802-4. Epub 2024 Feb 6. PMID 38321220